CLINICAL TRIAL: NCT06690333
Title: Efficacy and Safety of Leadless Pacemakers Versus Left Bundle Area Pacing - A Preliminary Exploration
Acronym: COMPAREPACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NCH Healthcare System, Inc. dba Naples Comprehensive Health and dba NCH (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dinesh Sharma, MD, NCH Healthcare System, Inc. dba Naples Comprehensive Health and dba NCH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB0081; 13500 (Other: Medtronic)
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pacemaker Implantation; AV Node Disease
Keywords: pacemaker; MICRA AV; Leadless pacemaker; left bundle area pacing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical Events Committee is masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Left bundle area pacing (Active Comparator): Transvenous pacemaker with left bundle area pacing
  Interventions: Device: Pacemaker
- MICRA AV (Active Comparator): Transcatheter pacemaker with MICRA AV
  Interventions: Device: Pacemaker

INTERVENTIONS:
Device: Pacemaker — Transvenous pacemaker with left bundle area pacing
  Arms: Left bundle area pacing
Device: Pacemaker — Transcatheter pacemaker with MICRA AV
  Arms: MICRA AV

SUMMARY:
This is a prospective, randomized controlled (1:1) multicenter trial. The pilot study will be conducted up to three clinical sites in the United States. The primary purpose of this study is to compare the overall safety and efficacy between the leadless pacemaker and left bundle area pacing.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled (1:1) multicenter trial. The pilot study will be conducted up to three clinical sites in the United States. This study is designed to compare the safety and effectiveness of two types of pacemaker treatments: leadless pacemakers and left bundle area pacing. Patients who's heart rhythm indicate a degree of heart block that slows the heart beat and decreases the amount of blood the heart is pumping to the rest of the body will be identified by physicians to participate. This study seeks to improve our understanding of heart rhythm disorders to allow us to provide the best treatment for our patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Planned for:

   1. permanent pacemaker implantation for AV node disease (first, second or third degree), OR
   2. post-TAVR patient requiring permanent pacemaker implantation
3. Preserved ejection fraction > 50%
4. Preserved sinus node function
5. Willingness to adhere to study restrictions and comply with all post-procedural follow-up requirements
6. Life expectancy > 1 year
7. Female subject of childbearing potential is not pregnant, not breast feeding, does not plan to be pregnant during the course of the study, and agrees to use a highly effective contraceptive method (i.e. IUD, birth control, vasectomized partner, sexual abstinence, etc.) during the course of the study.
8. Subject has been informed of the nature of the study, agrees to its provision and has provided written informed consent, approved by the IRB

Exclusion Criteria:

1. Sinus node dysfunction, anticipating atrial pacing or persistent atrial fibrillation
2. Anatomical restriction for either MICRA or transvenous pacing such as

   1. Access vein occlusion or thrombosis
   2. previous radiation therapy at insertion site
   3. inferior vena cava filter
3. Endstage renal disease (ESRD)/on dialysis
4. Dementia (inability to give consent)
5. Moderate to Severe or Severe Tricuspid valve regurgitation
6. Moderate to Severe or Severe Mitral valve regurgitation
7. History of mitral or tricuspid valve surgery
8. Preexisting implanted pacemaker or ICD or lead
9. Subject is allergic to titanium
10. Life expectancy < 1 year
11. Recurrent or high risk of infections
12. Active malignancy requiring systemic chemotherapy or local chest radiation
13. Subject has myocardial infarction, unstable angina, cerebrovascular accident, or heart failure admission within 3 months of the baseline visit
14. CABG, valve surgery or PCI within the last 3 months except TAVR
15. Other major cardiac surgery within the last 6 months
16. Persistent and permanent atrial fibrillation diagnosed by a healthcare provider
17. NYHA class 3 or 4 Heart Failure

    Additional post-TAVR Exclusion Criteria:
18. Evidence of renal injury (12 hours post-TAVR)
19. Access site complication(s) post-TAVR
20. Suspicion of stroke/cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 12 hours post-TAVR
21. Physician suspicion that ambulation to pre-TAVR activities post-pacemaker implantation would be unattainable
22. Other post-TAVR complications that in the opinion of the investigator may seriously confound study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy & Safety | 12 months
  The composite of:
  1. procedural success
  2. freedom from serious device-related complications at one year
  3. freedom from heart failure or drop in ejection fraction below 50%.

SECONDARY OUTCOMES:
Procedure time | from procedure start to procedure end
  measured in minutes
Device longevity | at 12 month follow up
  device longevity as noted on interrogation reports

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Sharma, MD, Principal Investigator — NCH Healthcare
Locations (2):
- United States (2):
  - NCH Healthcare, Naples, Florida
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vijayaraman P, Sharma PS, Cano O, Ponnusamy SS, Herweg B, Zanon F, Jastrzebski M, Zou J, Chelu MG, Vernooy K, Whinnett ZI, Nair GM, Molina-Lerma M, Curila K, Zalavadia D, Haseeb A, Dye C, Vipparthy SC, Brunetti R, Moskal P, Ross A, van Stipdonk A, George J, Qadeer YK, Mumtaz M, Kolominsky J, Zahra SA, Golian M, Marcantoni L, Subzposh FA, Ellenbogen KA. Comparison of Left Bundle Branch Area Pacing and Biventricular Pacing in Candidates for Resynchronization Therapy. J Am Coll Cardiol. 2023 Jul 18;82(3):228-241. doi: 10.1016/j.jacc.2023.05.006. Epub 2023 May 21. PMID 37220862
- [Background] Chinitz L, Ritter P, Khelae SK, Iacopino S, Garweg C, Grazia-Bongiorni M, Neuzil P, Johansen JB, Mont L, Gonzalez E, Sagi V, Duray GZ, Clementy N, Sheldon T, Splett V, Stromberg K, Wood N, Steinwender C. Accelerometer-based atrioventricular synchronous pacing with a ventricular leadless pacemaker: Results from the Micra atrioventricular feasibility studies. Heart Rhythm. 2018 Sep;15(9):1363-1371. doi: 10.1016/j.hrthm.2018.05.004. Epub 2018 May 11. PMID 29758405
- [Background] Sanchez R, Nadkarni A, Buck B, Daoud G, Koppert T, Okabe T, Houmsse M, Weiss R, Augostini R, Hummel JD, Kalbfleisch S, Daoud EG, Afzal MR. Incidence of pacing-induced cardiomyopathy in pacemaker-dependent patients is lower with leadless pacemakers compared to transvenous pacemakers. J Cardiovasc Electrophysiol. 2021 Feb;32(2):477-483. doi: 10.1111/jce.14814. Epub 2020 Nov 25. PMID 33205561
- [Background] Duray GZ, Ritter P, El-Chami M, Narasimhan C, Omar R, Tolosana JM, Zhang S, Soejima K, Steinwender C, Rapallini L, Cicic A, Fagan DH, Liu S, Reynolds D; Micra Transcatheter Pacing Study Group. Long-term performance of a transcatheter pacing system: 12-Month results from the Micra Transcatheter Pacing Study. Heart Rhythm. 2017 May;14(5):702-709. doi: 10.1016/j.hrthm.2017.01.035. Epub 2017 Feb 10. PMID 28192207
- [Background] Udo EO, Zuithoff NP, van Hemel NM, de Cock CC, Hendriks T, Doevendans PA, Moons KG. Incidence and predictors of short- and long-term complications in pacemaker therapy: the FOLLOWPACE study. Heart Rhythm. 2012 May;9(5):728-35. doi: 10.1016/j.hrthm.2011.12.014. Epub 2011 Dec 17. PMID 22182495
- [Background] Vijayaraman P, Ponnusamy S, Cano O, Sharma PS, Naperkowski A, Subsposh FA, Moskal P, Bednarek A, Dal Forno AR, Young W, Nanda S, Beer D, Herweg B, Jastrzebski M. Left Bundle Branch Area Pacing for Cardiac Resynchronization Therapy: Results From the International LBBAP Collaborative Study Group. JACC Clin Electrophysiol. 2021 Feb;7(2):135-147. doi: 10.1016/j.jacep.2020.08.015. Epub 2020 Oct 28. PMID 33602393
- [Background] Zhang S, Guo J, Tao A, Zhang B, Bao Z, Zhang G. Clinical outcomes of left bundle branch pacing compared to right ventricular apical pacing in patients with atrioventricular block. Clin Cardiol. 2021 Apr;44(4):481-487. doi: 10.1002/clc.23513. Epub 2021 Mar 11. PMID 33704810
- [Background] Kiehl EL, Makki T, Kumar R, Gumber D, Kwon DH, Rickard JW, Kanj M, Wazni OM, Saliba WI, Varma N, Wilkoff BL, Cantillon DJ. Incidence and predictors of right ventricular pacing-induced cardiomyopathy in patients with complete atrioventricular block and preserved left ventricular systolic function. Heart Rhythm. 2016 Dec;13(12):2272-2278. doi: 10.1016/j.hrthm.2016.09.027. PMID 27855853
- [Background] Kusumoto FM, Schoenfeld MH, Barrett C, Edgerton JR, Ellenbogen KA, Gold MR, Goldschlager NF, Hamilton RM, Joglar JA, Kim RJ, Lee R, Marine JE, McLeod CJ, Oken KR, Patton KK, Pellegrini CN, Selzman KA, Thompson A, Varosy PD. 2018 ACC/AHA/HRS Guideline on the Evaluation and Management of Patients With Bradycardia and Cardiac Conduction Delay: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Circulation. 2019 Aug 20;140(8):e382-e482. doi: 10.1161/CIR.0000000000000628. Epub 2018 Nov 6. No abstract available. PMID 30586772
- [Background] Huang HD, Mansour M. Pacemaker Implantation After Transcatheter Aortic Valve Replacement: A Necessary Evil Perhaps But Are We Making Progress? J Am Heart Assoc. 2020 May 5;9(9):e016700. doi: 10.1161/JAHA.120.016700. Epub 2020 May 2. No abstract available. PMID 32362173
- [Background] Dell'Era G, Baroni M, Frontera A, Ghiglieno C, Carbonaro M, Penela D, Romano C, Giordano F, Del Monaco G, Galimberti P, Mazzone P, Patti G. Left bundle branch area versus conventional pacing after transcatheter valve implant for aortic stenosis: the LATVIA study. J Cardiovasc Med (Hagerstown). 2024 Jun 1;25(6):450-456. doi: 10.2459/JCM.0000000000001619. Epub 2024 Apr 1. PMID 38625833
- [Background] Kassab K, Patel J, Feseha H, Kaynak E. MICRA AV implantation after transcatheter aortic valve replacement. Cardiovasc Revasc Med. 2024 Jun;63:31-35. doi: 10.1016/j.carrev.2024.01.005. Epub 2024 Jan 12. PMID 38220556
- [Background] Mechulan A, Prevot S, Peret A, Nait-Saidi L, Miliani I, Leong-Feng L, Leude-Vaillant E, Vaillant A, Cornen A, Latiere B, Giacomoni MP, Collet F, Bechet V, Bouharaoua A, Dieuzaide P. Micra AV leadless pacemaker implantation after transcatheter aortic valve implantation. Pacing Clin Electrophysiol. 2022 Nov;45(11):1310-1315. doi: 10.1111/pace.14545. Epub 2022 Jun 13. PMID 35661380